CLINICAL TRIAL: NCT01059383
Title: Active Control, Double-blind, Double-dummy, Parallel-group, Randomized Study to Assess the Effect of VECAM 40/300, Administered at Bedtime, vs. Esomeprazole 20 mg, Administered 30-60 Min. Before Dinner, on Daytime and Nighttime GERD Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vecta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCT007
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; GERD; Nocturnal GERD; Heartburn; Nighttime Heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- VECAM 40/300 (Experimental)
  Interventions: Drug: VECAM 40/300
- Esomeprazole 20 mg (Active Comparator)
  Interventions: Drug: Esomeprazole 20 mg

INTERVENTIONS:
Drug: VECAM 40/300 — 1 capsule, orally, once daily at bedtime.
  Arms: VECAM 40/300
Drug: Esomeprazole 20 mg — 1 capsule, orally, once daily 30-60 min. before dinner
  Arms: Esomeprazole 20 mg

SUMMARY:
The study is designed to assess the effect and safety of oral administration of VECAM 40/300 administered at bedtime compared to Esomeprazole 20 mg administered 30-60 minutes before dinner, for control of nighttime and daytime HB and other 24 hour GERD symptoms.

The rational for the study is based on the contention that VECAM exhibits potent inhibition of acid secretion and because of its mechanism of action, it can be administered at bedtime without food. Such timing of drug dosing will allow effective inhibition of nighttime acid secretion. Because of its mechanism of action, VECAM exhibits improved 24-hour inhibition of acid secretion and hence, its bedtime administration will not compromise its effect during the daytime. This improved control of acid secretion will predictably result in better control of nighttime as well as daytime heartburn (HB) symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Male or female
* H. pylori negative status
* Suffering from nighttime and daytime heartburn for the last ≥3 months
* At least 28 days of PPI use prior to study entry
* Patients have to be current PPI users with either:

  * Category 1): ≥ 2 HB episodes in 7 consecutive days, at least one during the nighttime to approved PPI doses, or
  * Category 2): only obtaining complete relief of GERD symptoms following the addition of acid suppressive agents (e.g. H2RA, additional PPI dose), or antacid therapy, to the approved PPI dose.
* Reporting of ≥ 3 HB episodes in 7 consecutive days, at least two during the nighttime, w/o medical treatment during a screening period of up to 21 days (report is based on a daily diary during the screening period) and for Category 1 patients, at least one more HB episode as compared to single dose treatment period.
* Use of acceptable form of birth control in females with child-bearing potential
* Can swallow a size "00" capsule without difficulty
* Willing to comply with study protocol
* Understood and signed an informed consent form for this study

Exclusion Criteria:

* BMI > 40
* Slow or poor Omeprazole metabolizers (heterozygous or homozygous, respectively based on CYP2C19 genotyping test.
* Any significant history of / or concurrent gastrointestinal diseases or conditions including:
* Acute gastrointestinal bleeding. or history of GI bleeding within 6 months prior to randomization
* Zollinger Ellison Syndrome or Gastric hypersecretory condition
* Esophageal stricture
* Active gastric or duodenal ulcers within 30 days prior to randomization
* Gastric outlet obstruction
* Gastro-paresis or gastric emptying disorder
* Significant hepatic disease: cirrhosis or hepatic encephalopathy
* Any significant medical co-morbidity that precludes participation in the study or can affect acid secretion, or sleep as judged by the investigator
* Significant laboratory abnormalities as determined by the principal investigator.
* Known metabolic alkalosis, hypocalcemia, sodium restricted diet, hypokalemia, or respiratory alkalosis.
* Had been treated with any investigational drug or therapy or participated in a clinical trial within 30 days prior to entering the trial.
* Active or illicit drug or alcohol abuse
* Use of any medication that alters gastric acid secretion other than the study medications provided by the study personnel.
* Regular use (>3 doses per week) of non-steroidal anti-inflammatory drugs (NSAIDs), including COX 2 inhibitors within 30 days prior to randomization or during the study.
* Use of the following medications during the study:

  * Bismuth-containing products
  * Antibiotics
  * Sucralfate
  * Misoprostol
  * Corticosteroids
  * Prokinetic agents
  * Anticoagulant therapy
  * Antiseizure medications
  * Psychotropic medications
  * Narcotic medications
  * Bisphosphonates
  * Anti-neoplastic treatments
  * Use of sleep medications:
  * First generation antihistamines
  * Benzodiazepines
  * Modified cyclic antidepressants
  * Antianxiety medications
  * Unless dose remains unchanged throughout the study, drugs with significant anticholinergic effects such as tricyclic antidepressants or drugs with CNS effects that could mask perception of symptoms (e.g., SSRIs*, SNRIs**).
  * Unless consumed during the screening period per protocol instructions:
  * Proton pump inhibitors (other than the study medication)
  * Histamine (H2) receptor antagonists
* Any conditions other than GERD that could be the primary cause of significant sleep disturbances (including but not limited to anxiety, depression, panic attacks, sleep apnea, chronic obstructive pulmonary disease requiring oxygen therapy or that are known to disrupt patients sleep, chronic insomnia, excessive use of caffeine), nocturnal urination
* Pregnant or lactating women
* Had been treated with any investigational drug or therapy or participated in a clinical trial within 30 days prior to entering the trial
* Significant drug allergy or known hypersensitivity to: any proton pump inhibitor drug , or ingredients in the study medications (Omeprazole, Succinic Acid) or their inactive ingredients contained in their capsule, or to Gelusil® tablets
* Had donated blood within 30 days of entering the trial
* Known positive serology for HBV, HCV or HIV
* Diabetes
* Any reason that makes the patient a poor candidate based on the study physician, or PI's discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Percentage of days with neither daytime nor nighttime heartburn during week 1, 2, 3, 4 and the overall treatment period measured with a patient-reported HB daily diary | 4 weeks

SECONDARY OUTCOMES:
Complete resolution of nighttime and daytime HB during the subject's last 7 diary reported days in the study, | 4 weeks
Percentage of days without nighttime HB on week 1, 2, 3, 4 and the overall treatment period, measured with a patient-reported HB daily diary. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Applications Laboratories Inc., San Diego, California
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma